CLINICAL TRIAL: NCT06051747
Title: Development of the Practical Usage Based Technology Using the Patient Customized Bioprinting Trachea for the Regeneration of Respiratory Tract (Trachea)
Brief Title: Patient-Customized Bioprinting Technology for Practical Regeneration of the Respiratory Tract (Trachea)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ja Seong Bae, MD, phD (Other)
Collaborators: Korea Health Industry Development Institute (Other Government)
Responsible Party: Sponsor-Investigator, Ja Seong Bae, MD, phD, Professor, Seoul St. Mary's Hospital
Organization: Seoul St. Mary's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMCENT-02
Record Dates: First submitted 2023-08-29; First posted 2023-09-25 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Thyroid Cancer
Keywords: Trachea
MeSH Terms: conditions — Thyroid Neoplasms; Tracheal Diseases

STUDY DESIGN:
Intervention Model Description: Treatment group : 1 patient with bioprinted tracheal reconstruction
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treated (Experimental): Three-dimensional patient-specific bioprinting trachea implantation
  Interventions: Procedure: Three-dimensional patient-specific bioprinting trachea implantation

INTERVENTIONS:
Procedure: Three-dimensional patient-specific bioprinting trachea implantation — The intervention entails the creation of a 3D cell-printed tracheal organ, achieved through the fusion of biopolymer materials and the bioprinting (3D cell printing) technique. This process involves distribution of nasal cavity stem cells (hNTSCs) and nasal septum cartilage cells (hNCs) within hydrogel matrices, culminating in the formation of a personalized tracheal structure.

SUMMARY:
This clinical trial aims to assess the effectiveness and safety of a novel approach utilizing biopolymers, hydrogels, mucous membranes, and cartilage tissue regeneration cells integrated into 3D bioprinting technology for the creation and implantation of patient-specific tracheal organs.

DETAILED DESCRIPTION:
Study Objective:

This clinical study focuses on patients with thyroid or airway diseases necessitating partial or segmental organ resection. The objective is to evaluate the feasibility, efficacy, and safety of transplanting functional patient-specific bioprinted tracheal organs as an innovative regenerative approach.

Patient Enrollment:

Patients voluntarily participate and provide written consent. A thorough screening procedure is conducted to determine their eligibility based on selection and exclusion criteria.

Bioprinting Process:

The study employs cutting-edge bioprinting technology to create complex organ tissues. Specifically, 3D cell printing is employed to fabricate a bioprinted tracheal organ. Stem cells derived from the human nasal cavity and nasal septum cartilage cells are integrated to form a cell-supporting body.

Transplantation Procedure:

Eligible patients receive transplantation of the functional patient-specific bioprinted trachea. The transplantation aims to restore tracheal functionality and address the unique challenges posed by thyroid and airway diseases.

Evaluation and Monitoring:

Following transplantation, a comprehensive assessment regimen is undertaken to evaluate both the effectiveness and safety of the procedure. This includes flexural laryngeal endoscopy, bronchoscopy, computed tomography (CT) scans, and laboratory tests.

Post-Transplant Measures:

To ensure the stability of the transplanted organ immediately after the procedure, neck fixing splints are employed to limit movement.

Thyroid Cancer Patients:

For patients diagnosed with thyroid cancer, a distinct follow-up protocol is established. A five-year observation period is implemented, extending beyond the standard follow-up for general cancer patients. Additional observations include thyroid ultrasound, Free T4, Thyroid-Stimulating Hormone (TSH), Thyroglobulin Antigen (Thyroglobulin Ag), and Anti-Thyroglobulin Antibody (Anti-TG Ab) tests conducted at the designated observation points.

This study seeks to contribute novel insights into the realm of regenerative medicine and enhance the understanding of patient-specific bioprinting technology as a potential solution for tracheal and airway diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Age Range:

   Individuals between 19 and 75 years of age are eligible for participation.
2. Specific Medical Condition:

   Patients must meet the following criteria and have thyroid or airway diseases necessitating partial or segmental resection:
   1. Thyroid Cancer Patients:

      For patients with thyroid cancer, inclusion is based on TNM staging, specifically stage II or higher differentiated thyroid cancer patients. Verification of complete removal through a freeze section test during surgery in accordance with the staging system for papillary carcinoma of the trachea is essential (Hum Pathol. 1993 Aug; 24(8):866-70).

      Patients for whom conventional reconstruction methods, including single-stage anastomosis, are infeasible and require alternative approaches like flap reconstruction.

      Patients suitable for single anastomosis, but assessed to derive more benefits than risks from 3D bioprinting, considering factors such as post-surgery aftereffects, complications, prolonged recovery, and potential decline in quality of life due to surgical intervention.
   2. Defect Size Patients with defects encompassing more than 30% of the cartilage around the affected organ are eligible. Smaller defects may also qualify if reinforcing defects using soft tissue is infeasible due to factors such as surrounding inflammation, tissue instability, tissue adhesion, unstable blood supply, or the anticipation of reoperation during reconstruction.
3. Pregnancy Consideration:

   In the case of childbearing women, individuals must provide a negative result on a pregnancy test and commit to using contraception throughout the clinical study period.
4. Informed Consent:

Participants must voluntarily provide written consent after receiving a comprehensive explanation of the clinical study.

Exclusion Criteria:

1. Pregnancy and Lactation:

   Pregnant or lactating women are excluded from participation in the study.
2. Prior Thyroid or Airway Surgery:

   Individuals who have undergone thyroid or airway peripheral surgery before undergoing screening are ineligible for participation.
3. Persistent Inflammation:

   Patients with ongoing inflammation of the thyroid or surrounding tissues at the time of screening are excluded.
4. Systemic Inflammatory Disease:

   Patients diagnosed with systemic inflammatory diseases at the screening stage are not eligible to participate.
5. Anesthesia Risk Factors:

   Individuals with a high risk of complications associated with general anesthesia due to existing liver disease, kidney disease, or heart disease are excluded.
6. Sepsis:

   Patients diagnosed with sepsis at the time of screening are not eligible for participation.
7. Hemorrhage Predisposition:

Individuals with a predisposition to hemorrhage at the time of screening are excluded from the study.

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2025-08-16 (Estimated)

PRIMARY OUTCOMES:
airway lumen opening rate | 1 week, 2 weeks, 4 weeks, 24 weeks, 2 years
  measured by curved laryngeal endoscopy
crust formation degree | 1 week, 2 weeks, 4 weeks, 24 weeks, 2 years
  measured by curved laryngeal endoscopy
granuloma formation degree | 1 week, 2 weeks, 4 weeks, 24 weeks, 2 years
  measured by curved laryngeal endoscopy
degree of inflammation | 1 week, 2 weeks, 4 weeks, 24 weeks, 2 years
  measured by curved laryngeal endoscopy
other relevant findings | 1 week, 2 weeks, 4 weeks, 24 weeks, 2 years
  measured by curved laryngeal endoscopy

SECONDARY OUTCOMES:
Airway State on CT | 4 weeks
  airway patency by ratio compared to preoperative state
white blood cell count (WBC) | 4 weeks, 48 weeks, 2years
  Serum inflammatory markers
differential white blood cell count (WBC Diff) | 4 weeks, 48 weeks, 2years
  Serum inflammatory markers
C-reactive protein (CRP) | 4 weeks, 48 weeks, 2years
  Serum inflammatory markers
erythrocyte sedimentation rate (ESR) | 4 weeks, 48 weeks, 2years
  Serum inflammatory markers
stability of bronchial wall structure | 4 weeks, 48 weeks, 2years
  measured by bronchoscopy
degree of organ opening | 4 weeks, 48 weeks, 2years
  measured by bronchoscopy
mucous membrane formation | 4 weeks, 48 weeks, 2years
  measured by bronchoscopy
presence of inflammatory or healing tissue | 4 weeks, 48 weeks, 2years
  measured by bronchoscopy

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 1 week, 2 weeks, 4 weeks, 24 weeks, 48 weeks, 72 weeks, 2 years
  Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Sung Won Kim, MD, PhD, Study Chair — Seoul St. Mary's Hospital
Locations (1):
- Seoul St. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Park JH, Hong JM, Ju YM, Jung JW, Kang HW, Lee SJ, Yoo JJ, Kim SW, Kim SH, Cho DW. A novel tissue-engineered trachea with a mechanical behavior similar to native trachea. Biomaterials. 2015 Sep;62:106-15. doi: 10.1016/j.biomaterials.2015.05.008. Epub 2015 May 23. PMID 26041482
- [Result] Park JH, Park JY, Nam IC, Ahn M, Lee JY, Choi SH, Kim SW, Cho DW. A rational tissue engineering strategy based on three-dimensional (3D) printing for extensive circumferential tracheal reconstruction. Biomaterials. 2018 Dec;185:276-283. doi: 10.1016/j.biomaterials.2018.09.031. Epub 2018 Sep 19. PMID 30261427
- [Result] Park JH, Park JY, Nam IC, Hwang SH, Kim CS, Jung JW, Jang J, Lee H, Choi Y, Park SH, Kim SW, Cho DW. Human turbinate mesenchymal stromal cell sheets with bellows graft for rapid tracheal epithelial regeneration. Acta Biomater. 2015 Oct;25:56-64. doi: 10.1016/j.actbio.2015.07.014. Epub 2015 Jul 9. PMID 26163763

DOCUMENTS (2):
  • Study Protocol (2023-05-26): https://cdn.clinicaltrials.gov/large-docs/47/NCT06051747/Prot_000.pdf
  • Informed Consent Form (2023-07-19): https://cdn.clinicaltrials.gov/large-docs/47/NCT06051747/ICF_001.pdf